CLINICAL TRIAL: NCT01185483
Title: Endoscopic Submucosal Dissection in Upper Gastrointestinal Canal With HybridKnife
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Michael Bau Mortensen, Odense University Hospital
Other Study IDs: ESD-HYBRID-AFDA
Record Dates: First submitted 2010-08-17; First posted 2010-08-20 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-08

CONDITIONS: Endoscopy, Digestive System; Esophageal Neoplasms; Stomach Neoplasms
Keywords: Endoscopic submucosal dissection; Submucosal tumor; Minimal invasive; Gastroscopy
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Endoscopic submucosal dissection (ESD) is a relatively new modality for the treatment of superficial gastrointestinal neoplasia and especially in the diagnosis and treatment of submucosal tumors. ESD has become a minimal invasive alternative to surgery but requires a high degree of endoscopic skills to be performed safely, it is time consuming, and less safe than endoscopic mucosa resection.

New endoscopic instruments have been developed to increase the efficacy and safety of ESD, and a combined endoscopic instrument (HybridKnife) has been developed and evaluated with promising results in animal studies. This HybridKnife allows high-pressure water-jet (submucosal) dissection, as well as cutting and coagulation and makes ESD possible without changing instrument.

The purpose of this study is to evaluate the feasibility and safety of using HybridKnife for ESD in humans.

ELIGIBILITY:
Inclusion Criteria:

* Submucosal tumor (< 4 cm)
* Mucosal tumor (T1) in patients unsuitable for surgery

Exclusion Criteria:

* Endoscopic ultrasound (EUS) or CT signs of metastasis
* Insufficient access to tumor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Endoscopic Section at the Department of Surgery, Odense University Hospital, with a mucosal or submucosal tumor in the esophagus or stomach.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Estimated); Study Completion 2011-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark